CLINICAL TRIAL: NCT06479161
Title: Effects of Oral Tranexamic Acid Following Total Knee Arthroplasty on Postoperative Pain and Range of Motion: A Randomized Control Trial
Brief Title: Effects of Oral Tranexamic Acid Following Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Grosso, MD (Other)
Responsible Party: Sponsor-Investigator, Matthew Grosso, MD, Director, Quality and Outcomes Research, Trinity Health Of New England
Organization: Trinity Health Of New England (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFH 24-05
Record Dates: First submitted 2024-06-20; First posted 2024-06-28 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This will be a double blinded study, with both patient and surgeon blinded to study group.
  Collaboration with Saint Francis' pharmacy team will be performed to ensure appropriate blinded administering of the oral TXA and placebo medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TXA (Active Comparator): - 1.95 grams oral TXA (tranexamic acid) (3- 650 mg tablets) administered postop day one, postop day two and postop day three. Compounded by registered pharmacist and labeled with subject name and instructions for use.
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): - 3 tablets administered postop day one, postop day two and postop day three. Compounded by registered pharmacist and labeled with subject name and instructions for use.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — 1.95 grams oral

SUMMARY:
The primary purpose of this study is to evaluate postoperative pain. Secondary outcomes evaluated in this study will include range of motion (ROM), opioid consumption, and ambulation. Each outcome measure will be evaluated, oral tranexamic acid (TXA) in the experiment arm and placebo in the control arm, after total knee arthroplasty (TKA) at postoperative days 0-3, and weeks 1, 2, 6, and 12.

DETAILED DESCRIPTION:
Randomized controlled trial with 1:1 allocation, selected through computer-based randomization.

This study will review prospectively collected data, including patient demographic information, surgeon, use of oral tranexamic acid (TXA) or placebo regimen, and postoperative outcomes up to 3 months after surgery. Collaboration with Saint Francis' pharmacy team will be performed to ensure appropriate blinded administering of the oral TXA and placebo medication.

This will be a double blinded study, with both patient and surgeon blinded to study group.

6.0 TXA dosing protocol TXA day of surgery [All patients]

* Administer 1-gram IV TXA intraoperatively at the start of the case (hold for history of stent within 1 year of surgery)

  o AND
* Administer 1-gram IV TXA postoperatively before leaving PACU (hold for history of stent within 1 year of surgery)

  o OR
* Exception: Administer 2 grams TXA in 50cc normal saline topically during the case for patients with a history of stent placed within one year of surgery.

TXA postoperative day (POD) 1-3 [Experimental group]

* Administer 1.95 grams oral (3- 650 mg tablets) TXA each morning for three days following surgery.
* Patients discharged home before POD 3 will be sent home with remaining oral TXA doses.

Placebo POD 1-3 [Control group]

* Administer oral placebo (3 tablets) each morning for three days following surgery.
* Patients discharged home before POD 3 will be sent home with remaining oral placebo doses.

ELIGIBILITY:
Inclusion Criteria:

* - All patients undergoing either manual or robotic primary total knee arthroplasty (TKA)
* Performed by participating Connecticut Joint Replacement Institute (CJRI) surgeons (Dr. Matthew Grosso, Dr. Robert McAllister, Dr. Chad Daniel, Dr. Eric Silverstein, Dr. Alex Dukas, Dr. Michael Joyce, Dr. Brett Wasserlauf).
* Male and female patient age 18-89
* Primary diagnosis of knee osteoarthritis

Exclusion Criteria:

* Revision TKA
* No exclusion based on gender
* Patients <18 and >89 years old
* Exclusion for IV oral tranexamic acid (TXA):

  * TXA allergy - there are NO absolute contraindications for TXA use.
  * History of stent placed within one year of surgery - patient will receive topical TXA as an alternative.
* Exclusion for oral TXA:

  o Actively treated cancer or deep vein thrombosis (DVT)
* Chronic opioid use (opioid use within the 4 weeks prior to surgery)
* Allergies to nonsteroidal Anti-inflammatory drugs (NSAIDs) and acetaminophen
* Patients with clinically significant drug interactions
* Pre-existing neuropathy
* Current or previous venous thrombosis (DVT or venous stasis disease)
* Immuno-compromised secondary to medical condition
* Immune-suppressive medications, chemotherapy
* Pregnancy, breast feeding
* History of pain catastrophizing. Major depressive disorder
* History of suspected or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Currently on a neuroleptic agent [e.g., gabapentin, pregabalin (Lyrica), duloxetine (Cymbalta) etc.].
* Non-English speaking and reading patient populations
* Any clinically significant event or condition uncovered during the surgery (e.g., excessive bleeding, acute sepsis) that, in the opinion of the investigator, renders the subject medically unstable or complicates the subject's post-operative course.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Pain scores | postoperative day (POD) 0, 1, 2, 3 (+/- 0 days) and weeks 1 (+/- 0 days), 2 (+/- 2 days), 6 and 12 (+/- 7 days).
  Patient reported pain score from 0 to 10 where 0 is no pain and 10 is the most pain. Higher scores are a worse outcome.

SECONDARY OUTCOMES:
Range of Motion | at 2, 6 and 12 week follow up visits
  Clinical measurement of passive, pain-free range of motion of knee in degrees from 0 to 180 from maximum extension to maximum flexion
Opioid consumption | POD 1, 2, 3 (+/- 0 days) and weeks 1 (+/- 0 days), 2 (+/- 2 days), 6 and 12 (+/- 7 days)
  Subjects will keep a log recording opioid consumption. Research staff will ask subjects to report opioids during postoperative telephone calls.
Ambulation Status | at 2, 6 and 12 week follow up visits
  Surgeon or physical therapist will record if patient is using a walker, cane or no assistive devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Trinity Health Of New England/CT Joint Replacement Institute, Hartford, Connecticut, United States